CLINICAL TRIAL: NCT02661672
Title: INVEST-REGISTRY: Minimally Invasive Endoscopic Surgical Treatment With Apollo/Artemis in Patients With Brain Hemorrhage: A Prospective Multicenter Registry
Brief Title: INVEST-REGISTRY: Minimally Invasive Endoscopic Surgical Treatment With Apollo/Artemis in Patients With Brain Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J. Mocco (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); University at Buffalo (Other)
Responsible Party: Sponsor-Investigator, J. Mocco, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-0028
Record Dates: First submitted 2016-01-11; First posted 2016-01-22 (Estimated); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Intracranial Hemorrhage
Keywords: Intracranial hemorrhage; Neurosurgery
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Brain Hemorrhage (Experimental): Subjects will receive best medical management for ICH plus they will receive the MIES surgery and use of the Apollo or Artemis System for clot evacuation.
  Interventions: Device: Apollo Device; Device: Artemis Device

INTERVENTIONS:
Device: Apollo Device — The Apollo system has been cleared for the controlled aspiration of soft tissue and/or fluid during endoscopically guided neurosurgery of the ventricular system.
  Other Names: ICH - Apollo System
Device: Artemis Device — The Artemis Neuro Evacuation Device is used for the controlled aspiration of tissue and/or fluid during surgery of the Ventricular System or Cerebrum in conjunction with a Penumbra Aspiration Pump. The Penumbra Aspiration Pump is indicated as a vacuum source for the Penumbra Aspiration Systems.

SUMMARY:
Objective: The primary objective of this multicenter prospective registry is to provide additional safety, technical outcomes and clinical outcomes data for minimally invasive endoscopic surgery (MIES) with Apollo or Artemis for the evacuation of supratentorial brain hemorrhage in adult patients who do not qualify for the concurrent INVEST Feasibility randomized controlled trial at active INVEST centers.

DETAILED DESCRIPTION:
Study Design: This study will be a prospective, non-randomized, multi-center, single arm registry that will enroll up to 50 patients, however may increase to 200 at up to 10 US centers.

Patient Population: Adult patients with supratentorial brain hemorrhages (ICH and/or IVH) who do not meet all INCLUSION criteria or who meet one or more EXCLUSION criteria for the INVEST trial, but who will ultimately undergo MIES with Apollo or Artemis at active INVEST centers.

Indication: The Artemis Neuro Evacuation Device is used for the controlled aspiration of tissue and/or fluid during surgery of the Ventricular System or Cerebrum in conjunction with a Penumbra Aspiration Pump. The Penumbra Aspiration Pump is indicated as a vacuum source for the Penumbra Aspiration Systems. The Apollo system has been cleared for the controlled aspiration of soft tissue and/or fluid during endoscopically guided neurosurgery of the ventricular system. In the present study, the researchers propose to investigate the safety and efficacy of this system for the minimally invasive evacuation of brain hemorrhage - both IVH, IVH with ICH and ICH alone - in patients who do not qualify for the INVEST trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 022 years or older
* Supratentorial brain hemorrhage, which may be:

  1. Intracerebral (ICH)
  2. Primarily Intracerebral (ICH) with a component of intraventricular hemorrhage (IVH)
  3. Primarily intraventricular hemorrhage (IVH) with a component of ICH
  4. Intraventricular hemorrhage (IVH)
* Patient does not qualify for the concurrent INVEST Feasibility study

Exclusion Criteria:

* Imaging

  * Expanding hemorrhage on stability CT/MR scan
  * "Spot sign" identified on CTA (May perform a second CTA at 12 hours to demonstrate resolution)
  * Hemorrhagic lesion such as a vascular malformation (cavernous malformation, AVM etc), aneurysm, neoplasm
  * Hemorrhagic conversion of an underlying ischemic stroke
  * Infratentorial hemorrhage
  * Midbrain extension/involvement
* Coagulation Issues

  * Absolute and imminent (within 7 days of treatment) requirement for long-term, full-dose, anti-coagulation (e.g., Mechanical valve replacement (bio-prostatic valve is permitted), high risk atrial fibrillation)
  * Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
  * Uncorrected platelet count < 100 x 103 cells/mm3 or known platelet dysfunction
  * INR > 1.45, elevated prothrombin time or activated partial thromboplastin time (aPTT), which cannot be corrected or otherwise accounted for (i.e., lupus anti-coagulant)
* Patient Factors

  * High risk condition for ischemic stroke (high risk Afib (e.g., mitral stenosis with Afib), symptomatic carotid stenosis)
  * Requirement for emergent surgical decompression or uncontrolled ICP after EVD
  * Unable to obtain consent from patient or appropriate surrogate (for patients without competence)
  * Pregnancy, breast-feeding, or positive pregnancy test [either serum or urine] (Woman of child-bearing potential must have a negative pregnancy test prior to the study procedure.)
  * Evidence of active infection [indicated by fever (at or over 100.7 °F) and/or open draining wound] at the time of randomization
  * Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 180 days.
  * Based on investigator's judgment, patient does not have the necessary mental capacity to participate or is unwilling or unable to comply with protocol follow up appointment schedule.
  * Active drug or alcohol use or dependence that, in the opinion of the site investigator would interfere with adherence to study requirements.
  * Currently participating in another interventional (drug, device, etc) research project.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Mocco, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (7):
  - George Washington University, Washington D.C., District of Columbia
  - University of Louisville, Louisville, Kentucky
  - University of Buffalo, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Brain Hemorrhage
Started | 38
Completed | 33
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 63.5 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 15
  More than one race | 0
  Unknown or Not Reported | 3
Tobacco use [Count of Participants; unit: Participants]
  Never smoked | 23
  Previously smoked (quit > 6 months ago) | 6
  Currently smoking (or quit within the last 6 months) | 9
Cocaine or methamphetamine use [Count of Participants; unit: Participants] | 4
On anticoagulant therapy [Count of Participants; unit: Participants] | 6
On antiplatelet therapy [Count of Participants; unit: Participants] | 11
On NSAID therapy [Count of Participants; unit: Participants] | 0
On antihypertensive therapy [Count of Participants; unit: Participants] | 22
Medical comorbidities [Count of Participants; unit: Participants]
  Diabetes | 6
  Hypertension | 28
  Other cardiovascular disease | 0
Location of intracerebral hemorrhage [Count of Participants; unit: Participants]
  Deep | 18
  Lobar | 20
mRS before stroke [Count of Participants; unit: Participants] — modified Rankin Scale (mRS): 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  Participants
    0 | 30
    1 | 3
    2 | 2
    3 | 3
Intracerebral hemorrhage (ICH) volume [Median (Inter-Quartile Range); unit: milliliters] | 30.3 [17.7 to 48.8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Modified Rankin Score (mRS) ≤ 3 or mRS > 3
Description: Clinical Efficacy Endpoint: global disability assessed via the modified Rankin score (mRS). 180-day global disability assessed via the modified Rankin score (mRS), categorized as either mRS ≤ 3 or mRS > 3
Time Frame: 180 days
Population: one participant lost to follow-up after 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 37
Participants
  mRS ≤ 3 | 17
  mRS > 3 | 20

2. Primary Outcome: Number of Participants With Surgical Success Rate
Description: Technical Efficacy Endpoint measured by rate of surgical success. Surgical Success Rate is defined as reduction to < 15 cc total volume AND >60% reduction in hemorrhage volume on immediate post-treatment CT scan
Time Frame: immediately post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
Participants | 27

3. Primary Outcome: Number of Participants With Surgical Success Rate Regarding IVH
Description: Technical Efficacy Endpoint measured by rate of surgical success. Surgical Success Rate is defined as Intraventricular hemorrhage (IVH): mGraeb score of < 5 on day 7 CT scan
Time Frame: 7 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
Participants | 14

4. Primary Outcome: Rate of Mortality
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
Participants | 1

5. Secondary Outcome: Modified Rankin Score (mRS) at 30 Days
Description: 0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
Participants
  0 | 1
  1 | 2
  2 | 1
  3 | 6
  4 | 16
  5 | 7
  6 | 1
  Unavailable | 4

6. Secondary Outcome: Modified Rankin Score (mRS) at 90 Days
Description: as for outcome 5
Time Frame: 90 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
Participants
  0 | 2
  1 | 2
  2 | 5
  3 | 8
  4 | 6
  5 | 5
  6 | 2
  Unavailable | 8

7. Secondary Outcome: Length of Hospital Stay
Time Frame: average of 17 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
days | 14.5 [9.3 to 24.0]

8. Secondary Outcome: Number of Participants Requiring VPS
Description: Number of participants requiring Ventriculoperitoneal Shunt (VPS)
Time Frame: average of 17 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Brain Hemorrhage
Number analyzed (Participants) | 38
Participants | 3

ADVERSE EVENTS:
Time Frame: up to 6 months post-procedure
Arm/Group | Patients With Brain Hemorrhage
All-Cause Mortality (participants affected / at risk) | 4/38
Serious Adverse Events (participants affected / at risk) | 20/38
Other Adverse Events (participants affected / at risk) | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Brain Hemorrhage (N=38)
Abdominal pain (Gastrointestinal disorders) | 2
Acute hemorrhage (Nervous system disorders) | 1
Acute inflammatory demyelinating polyneuropathy (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration pneumonia/fever (Infections and infestations) | 1
C. diff infection (Infections and infestations) | 1
Cranioplasty infection (Infections and infestations) | 1
Deep venous thrombosis (Vascular disorders) | 2
Facial fractures (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
Deep seated right brain lesion due to brain abscess (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia (Infections and infestations) | 1
Polycythemia vera (Blood and lymphatic system disorders) | 1
Pulmonary embolism (Vascular disorders) | 2
R frontal ICH (Nervous system disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis secondary to aspiration (Infections and infestations) | 1
Stroke (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Wound infection and cerebral abscess (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Brain Hemorrhage (N=38)
Abdominal distension (Gastrointestinal disorders) | 1
Acute encephalopathy (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Aspiration pneumonia (Infections and infestations) | 1
Back rash (Immune system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Craniotomy site oozing (Injury, poisoning and procedural complications) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 4
Hematoma (Vascular disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Hyperchloremia (Investigations) | 1
Hypernatremia (Investigations) | 3
Hypertension/hypertensive episode (Vascular disorders) | 2
Hypomagnesemia (Investigations) | 1
Hypopotassemia (Investigations) | 1
Intraventricular hemorrhage (Nervous system disorders) | 1
L great toe abscess (Infections and infestations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Pulmonary edema (Reproductive system and breast disorders) | 1
Pulmonary emboli (Vascular disorders) | 1
Seizure (Nervous system disorders) | 2
Stroke (Nervous system disorders) | 2
Suicide attempt (Psychiatric disorders) | 1
Transaminitis (Investigations) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Worsening of chronic kidney disease (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT02661672/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT02661672/ICF_001.pdf